CLINICAL TRIAL: NCT03688009
Title: Brief Mindfulness-Based Family Psychoeducation Intervention for Chinese Students With Early Psychosis: A Mixed Methods Study
Brief Title: Mindfulness-Based Family Psychoeducation Intervention for Early Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 15604118
Record Dates: First submitted 2018-09-11; First posted 2018-09-27 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Psychotic Disorder
Keywords: mindfulness-based intervention; family psychoeducation; Chinese family caregivers; early psychosis; mixed methods design
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Family Psycho-Education (MBFBE) (Experimental): A programme focuses on non-judgmental attitudes, collaborative inquiry and self-care, including components of understanding early psychosis, medication, treatment management, mental health service collaboration, attention to caregiver's experiences and distress, strategies for improving communication and problem-solving, and crisis planning.
  Interventions: Behavioral: Mindfulness-Based Family Psycho-Education (MBFBE)
- Family Psycho-Education (FPE) (Active Comparator): A programme focuses on information giving, problem-solving and mutual support, including components of understanding early psychosis, medication, treatment management, mental health service collaboration, attention to caregiver's experiences and distress, strategies for improving communication and problem-solving, and crisis planning.
  Interventions: Behavioral: Family Psycho-Education (FPE)

INTERVENTIONS:
Behavioral: Mindfulness-Based Family Psycho-Education (MBFBE) — Six sessions includes: 1. Working with Caregiving Stress; 2. The Struggles of a Caregiver; 3. The Struggles of a Person in Recovery; 4. The Path of Recovery; 5. A Supportive Caregiving; and 6. Review of Learning.
  Arms: Mindfulness-Based Family Psycho-Education (MBFBE)
Behavioral: Family Psycho-Education (FPE) — Six sessions includes: 1. Working with Caregiving Stress; 2. The Struggles of a Caregiver; 3. The Struggles of a Person in Recovery; 4. The Path of Recovery; 5. A Supportive Caregiving; and 6. Review of Learning.
  Arms: Family Psycho-Education (FPE)

SUMMARY:
A brief Mindfulness-Based Family Psychoeducation programme is developed to reduce the caregiver's stress and to promote young people's recovery.

A randomized controlled trial will be conducted to compare a mindfulness-based family psychoeducation intervention, with an ordinary family psychoeducation intervention. 300 caregivers of a youth who have experienced early psychosis will be recruited.

Programme effectiveness will be assessed by comparing outcomes measuring caregiver's perceived stress, positive well-being, and the young people's mental health symptoms. As part of the programme activity, Photovoice approach is selected to explore the complex family experiences and the benefits of mindfulness from the caregiver's personal perspectives. Caregivers can offer their voices about their burdens, and how mindfulness can benefit to the families through their involvement in a photo taking activity during the psychoeducation programme.

DETAILED DESCRIPTION:
According to the World Health Organization Global Burden of Disease Study, for youth aged 10 to 24 years old, schizophrenia ranked as the third among all causes of disability. Schizophrenia shows a marked increase in prevalence after aged 15 and many manifests in early 20s. The term early psychosis is used for young people before and after their first identified psychotic episode.

The support of family members during the treatment and recovery of early psychosis is critical. Schizophrenia results in serious functional impairment, including a delimited social networks, termination or suspension of schooling. Caregivers encounter much psychological distress, particularly in handling the violent behaviours, suicidal ideation, failures in treatment, and other illness behaviours of such students. One-third of such caregivers have experienced emotional difficulties, such as depression. Family psychoeducation intervention has been recommended as a major component in the treatment of early psychosis.

International and local studies have reported positive outcomes using family psychoeducation interventions, but many limitations have also been identified. Many previous studies implemented an intensive programme design, with an emphasis on improvements in illness outcome of patients only. A recent review concluded that benefits of such programmes to caregivers were limited. There have been calls for a time-limited but more cost-effective programme for caregivers of a youth with early psychosis to mitigate the looming realities of eventual serious mental illness and family suffering. A brief Mindfulness-Based Family Psychoeducation programme is developed to reduce the caregiver's stress and to promote young people's recovery. Results from the pilot study suggested that such programme could reduce caregiver stress, and promote positive caregiving experience.

A more rigorous study is proposed using a mixed methods design. A randomized controlled trial will be conducted to compare a mindfulness-based family psychoeducation intervention, with an ordinary family psychoeducation intervention. 300 caregivers of a youth who have experienced early psychosis will be recruited, with the assistance of five NGO collaborators. Programme effectiveness will be assessed by comparing outcomes measuring caregiver's perceived stress, positive well-being, and the young people's mental health symptoms. As part of the programme activity, Photovoice approach is selected to explore the complex family experiences and the benefits of mindfulness from the caregiver's personal perspectives. Caregivers can offer their voices about their burdens, and how mindfulness can benefit to the families through their involvement in a photo taking activity during the psychoeducation programme.

ELIGIBILITY:
Inclusion Criteria:

* caregivers of a youth under the age of 35 and who has experienced EP, or has a diagnosis of SMI, in the last three years
* caregivers who have offered the care to the student for at least one year.

Exclusion Criteria:

* caregivers who have diagnoses of SMI or developmental disabilities, such as intellectual disabilities, which may present difficulties in comprehending the content of the programme.
* both caregivers and youth who refuse to receive regular psychiatric consultation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline caregiver's general stress level at 6 weeks and at 12 months | (1) Pretest baseline, (2) through intervention completion, 6 weeks, and (3) 12-month follow up after intervention completion
  Measured by Zarit Burden Interview (ZBI) (22 items) (Zarit, Reever, Bach-Peterson 1980), assessing caregivers' subjective burden. The total score ranges from 0 (low burden) to 88 (high burden).

SECONDARY OUTCOMES:
Change from baseline caregiver's caregiving experiences at 6 weeks and at 12 months | (1) Pretest baseline, (2) through intervention completion, 6 weeks, and (3) 12-month follow up after intervention completion
  Measured by Experience of Caregiving Inventory (Szmukler et al., 1996), with selected subscales of Stigma (5 items), Effects on the Family (7 items), Positive Experience in Caregiving (14 items), assessing caregivers' experience in the caregiving relationship.
  The Stigma score ranges from 0 (little experience of stigma) to 20 (much experience of stigma). The Effects on the Family score ranges from 0 (little negative effects on the family) to 28 (much negative effects on the family). The Positive Experience in Caregiving score ranges from 0 (little positive experience in caregiving) to 56 (much positive experience in caregiving).
  No total scores are calculated.
Change from baseline caregiver's physical health and mental health at 6 weeks and at 12 months | (1) Pretest baseline, (2) through intervention completion, 6 weeks, and (3) 12-month follow up after intervention completion
  Physical health measured by 14 item, Physical Distress subscale in Body-Mind-Spirit Well-Being Inventory (Ng et al., 2005), assessing caregivers' level of subjective distress caused by specific physical symptoms; mental health, i.e., Anxiety and Depression, measured by Hospital Anxiety and Depression Scale (Zigmond & Snaith, 1983), assessing caregivers' severity of anxiety and depression.
  The Physical Distress score ranges from 0 (low distress) to 140 (high distress). The Anxiety score ranges from 0 (low anxiety) to 21 (high anxiety). The Depression score ranges from 0 (low depression) to 21 (high depression).
  No total scores are calculated.
Change from baseline caregiver's well-being at 6 weeks and at 12 months | (1) Pretest baseline, (2) through intervention completion, 6 weeks, and (3) 12-month follow up after intervention completion
  Measured by WHO-5 Well-Being Index (Johansen, 1998), assessing caregivers' emotional well-being.
  The total score ranges from 0 (bad well-being) to 25 (good well-being).
Change from baseline caregiver's perceived family functioning at 6 weeks and at 12 months | (1) Pretest baseline, (2) through intervention completion, 6 weeks, and (3) 12-month follow up after intervention completion
  Measured by 5 item, Family APGAR Scale (Smilkstein, Ashworth, & Montano, 1982), with five subscales in adaptation, partnership, growth, affection and resolve, assessing parent's satisfaction of family functions.
  The total score ranges from 0 (dissatisfaction) to 10 (good satisfaction).
Change from baseline youth's recovery at 6 weeks and at 12 months | (1) Pretest baseline, (2) through intervention completion, 6 weeks, and (3) 12-month follow up after intervention completion
  Measured by Mental Health Recovery Measure (Young & Bullock, 2005), with 30 items in eight subscales relating to positive dimensions in recovery including Overcoming Stuckness (OS; 4 items), Self-Empowerment (SE; 4 items), Learning and Self-Redefinition (LSR; 4 items), Basic Functioning (BF; 4 items), Overall Well-Being (OWB; 4 items), New Potentials (NP; 4 items), Advocacy/Enrichment (A/E; 4 items) and Spirituality (2 items), assessing recovery-related experiences of people with severe mental illness.
  The total score ranges from 0 (bad recovery-related experiences) to 120 (good recovery-related experiences).
  OS, SE, LSR, BF, OWB, NP and A/E range from 0 (bad recovery-related experiences) to 16 (good recovery-related experiences).
  Spirituality ranges from 0 (bad recovery-related experiences) to 8 (good recovery-related experiences).
  Eight subscale scores are summed to compute a total score.
Change from baseline caregiver's interpersonal mindfulness at 6 weeks and at 12 months | (1) Pretest baseline, (2) through intervention completion, 6 weeks, and (3) 12-month follow up after intervention completion
  Measured by the Interpersonal mindfulness in Parenting Scale (Duncan, 2007), with 23 items in four factors in Compassion for Child (CC), Emotional Awareness in Parenting (EAP), Nonjudgmental Acceptance in Parenting (NAP) and Listening with Full Awareness (LFA) (Lo et al., 2018), assessing caregivers' quality of mindfulness specific to his or her family context.
  The total score ranges from 23 (low mindfulness) to 115 (high mindfulness). CC ranges from 7 (low compassion for child) to 35 (high compassion for child). EAP ranges from 6 (low emotional awareness in parenting) to 30 (high emotional awareness in parenting). NAP ranges from 6 (low nonjudgmental acceptance in parenting) to 30 (high nonjudgmental acceptance in parenting). LFA ranges from 4 (less likely listening with full awareness) to 20 (more likely listening with full awareness).
  Four subscale scores are summed to compute a total score.
Change from baseline caregiver's non-attachment at 6 weeks and at 12 months | (1) Pretest baseline, (2) through intervention completion, 6 weeks, and (3) 12-month follow up after intervention completion
  Measured by short form (8 items) of Non-attachment Scale (Sahdra, Shaver & Brown, 2010), assessing caregivers' subjective level of nonattachment.
  The total score ranges from 8 (low level of nonattachment) to 48 (high level of nonattachment).
Change from baseline youth's expressed emotion at 6 weeks and at 12 months | (1) Pretest baseline, (2) through intervention completion, 6 weeks, and (3) 12-month follow up after intervention completion
  Measured by 12 item Level of Expressed Emotion Scale (Cole & Kazarian, 1988), with subscales in Criticism (4 items), Hostility (4 items) and Over-Involvement (4 items), assessing patients' perceived expressed emotions from the most influential person.
  The total score ranges from 12 (low perceived expressed emotions) to 48 (high perceived expressed emotions).
  Criticism, Hostility and Over-Involvement scores range from 4 (low perceived expressed emotions from particular sources) to 16 (high perceived expressed emotions from particular sources).
  Three subscale scores are summed to compute a total score.
Change from baseline youth's psychiatric symptom at 6 weeks and at 12 months | (1) Pretest baseline, (2) through intervention completion, 6 weeks, and (3) 12-month follow up after intervention completion
  Measured by the Positive and Negative Syndrome Scale (PNSS) (Kay, Flszbein & Opler, 1988), subscales in Positive Scale (7 items), Negative Scale (7 items) and General Psychopathology Scale (16 items), assessing students' psychiatric symptoms.
  Positive Scale ranges from 7 (few positive syndromes) to 49 (many positive syndromes).
  Negative Scale ranges from 7 (few negative syndromes) to 49 (many negative syndromes).
  General Psychopathology Scale ranges from 16 (few general psychopathological symptoms) to 112 (many).
  No total scores are calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang ZJ, Lo HHM, Ho WC, Lau ENS, Ng SM, Mak WWS, Wong SYS, Hung KSY, Lai IYS, Lo CSL, Wong JOY, Lui SSY, Siu CMW, Yan EWC, Chan SHW, Lin E, Wong GOC, Mak JWH, Tam HSW, Tse IHH. Mindfulness-based family psychoeducation intervention for caregivers of young adults with first-episode psychosis: results at 9-month follow-up. Front Psychiatry. 2024 Sep 26;15:1460151. doi: 10.3389/fpsyt.2024.1460151. eCollection 2024. PMID 39391083
- [Derived] Zhang ZJ, Lo HHM, Ng SM, Mak WWS, Wong SYS, Hung KSY, Lo CSL, Wong JOY, Lui SSY, Lin E, Siu CMW, Yan EWC, Chan SHW, Yip A, Poon MF, Wong GOC, Mak JWH, Tam HSW, Tse IHH, Leung BFH. The Effects of a Mindfulness-Based Family Psychoeducation Intervention for the Caregivers of Young Adults with First-Episode Psychosis: A Randomized Controlled Trial. Int J Environ Res Public Health. 2023 Jan 5;20(2):1018. doi: 10.3390/ijerph20021018. PMID 36673773
- [Derived] Lo HH, Ho WC, Lau EN, Lo CW, Mak WWS, Ng SM, Wong SY, Wong JO, Lui SSY, Lo CS, Lin EC, Poon MF, Choi K, Leung CW. A Brief Mindfulness-Based Family Psychoeducation Intervention for Chinese Young Adults With First Episode Psychosis: A Study Protocol. Front Psychol. 2019 Mar 11;10:516. doi: 10.3389/fpsyg.2019.00516. eCollection 2019. PMID 30915004

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-17): https://cdn.clinicaltrials.gov/large-docs/09/NCT03688009/Prot_SAP_000.pdf